CLINICAL TRIAL: NCT04190485
Title: To Evaluate the Clinical Efficacy of the Probiotic Toothpastes in Patients With Moderate to Severe Gingivitis
Brief Title: To Evaluate the Efficacy of Probiotics Toothpastes in Improvement of Gingivitis and Prevention of Periodontal Diseases Via Modulating the Oral Microbiota
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GenMont Biotech Incorporation (Industry)
Collaborators: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: KMUHIRB-F(I)-20190123
Record Dates: First submitted 2019-12-03; First posted 2019-12-09 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Gingivitis
Keywords: Gingivitis; Probiotic; Toothpaste; Oral microbiota
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo and GMNL-143 Probiotic Toothpastes (Experimental): Subjects will receive placebo and GMNL-143 probiotic toothpastes.
  Interventions: Other: Placebo; Other: GMNL-143 Probiotic Toothpastes
- Placebo and GMNL-464 Probiotic Toothpastes (Experimental): Subjects will receive placebo and GMNL-464 probiotic toothpastes.
  Interventions: Other: Placebo; Other: GMNL-464 Probiotic Toothpastes

INTERVENTIONS:
Other: Placebo — Subjects will be randomized to one of two groups, using placebo toothpastes for 4 weeks, and then will enter a 1 week-washout and afterward will be crossed over to the opposite treatment for 4 weeks.
Other: GMNL-143 Probiotic Toothpastes — Subjects will be randomized to one of two groups, using GMNL-143 probiotic toothpastes toothpastes for 4 weeks, and then will enter a 1 week-washout and afterward will be crossed over to the opposite placebo for 4 weeks.
  Arms: Placebo and GMNL-143 Probiotic Toothpastes
Other: GMNL-464 Probiotic Toothpastes — Subjects will be randomized to one of two groups, using GMNL-464 probiotic toothpastes for 4 weeks, and then will enter a 1 week-washout and afterward will be crossed over to the opposite placebo for 4 weeks.
  Arms: Placebo and GMNL-464 Probiotic Toothpastes

SUMMARY:
Gingivalis is the one of the most common diseases of oral cavity, and affects more than 75% of adult populations worldwide. The present studies demonstrated that the addition of probiotics in toothpastes or mouthwashes could reduce dental plaques and gum inflammation, and improve oral health. This study was designed to assess the effectiveness of probiotic toothpastes during the supportive therapy of moderate to sever gingivalis patients.

DETAILED DESCRIPTION:
Previous studies have shown that probiotics could improve oral health including periodontal diseases, dental caries and halitosis via inhibiting periodontal pathogens, modulating periodontal microbiome, and regulating oral mucosal immunity. Heat-killed probiotics strain, Lactobacillus paracasei GMNL-143 or Lactobacillus rhamnosus GMNL-464 possessed great coaggregation abilities with oral pathogens and removed them after rinsing mouths. Besides, GMNL-143 can decrease the secretion of pro-inflammatory cytokines, increase the expression of anti-inflammatory cytokines, and inhibit the growth of dental pathogen Streptococcus mutans. Hence, it is suggested GMNL-143 or GMNL-464 probiotic toothpastes can ameliorate oral health of patients with gingivitis.

In this clinical study, the effectiveness of probiotic toothpastes during the supportive therapy of moderate to sever gingivalis patients will be clarified. A randomized, double-blind, crossover and placebo controlled clinical trial will be formed. This clinical trial will be conducted at Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung, Taiwan. 60 subjects with moderate to severe gingivitis will be enrolled. This trial will last for 9 weeks, starting from the time when the subjects begin to use probiotic toothpastes. Subjects who pass the screening phase will enter the first visit (week 0) and return in the 4th, 5th and 9th weeks. Subjects will be randomized to one of two groups, using probiotic toothpastes (GMNL-143 or GMNL-464) or placebo toothpastes to brush teeth for two minutes twice daily for 4 weeks, and then will enter a 1 week-washout and afterward will be crossed over to the opposite treatment for 4 weeks. Subjects will receive assessments of plaque index and gingivitis index, collection of samples including plaque, gingival cervical fluid and saliva, and questionnaires of oral health impact profile (OHIP) and gastrointestinal health at each visit.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects received a dental prophylaxis one week before enrollment.
2. Subjects in age of 20-59 years old.
3. Subjects are diagnosed with moderate to serve gingivitis. (Gingival index: 1.1-3.0)
4. Subjects have a minimum of 20 natural teeth.

Exclusion Criteria:

1. Subjects with immunodeficiency disease. (ex. HIV, Autoimmune disease…)
2. Subjects have severe dental caries or mucosal lesions in oral cavity.
3. Subjects who are undergoing orthodontic treatment.
4. Anti-inﬂammatory drugs or antibiotics therapy during this trial.
5. Pregnant and nursing women.
6. Smoking, alcohol or areca nut consumption.
7. Use of probiotic products (not including yogurt and yogurt drink) during this trial.
8. Use of mouthwash.
9. Participation in another clinical study.

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2022-05-13 (Actual); Study Completion 2022-05-13 (Actual)

PRIMARY OUTCOMES:
Gingival Index | 0, 4, 5, 9 weeks
  The gingivitis will be evaluated at baseline and different timepoint post-intervention by Gingival index. Gingival index for individual teeth= Total of gingival index of each tooth/No. of teeth present. The minimum score of TMQHPI is 0 (Normal gingival). The maximum score of TMQHPI is 3 (severe gingivitis).

SECONDARY OUTCOMES:
Plaque index | 0, 4, 5, 9 weeks
  The plaque accumulation will be evaluated by Turesky-Modified of the Quigley- Hein Plaque Index(TMQHPI) and plaque index at baseline and different timepoint post-intervention. TMQHPI Index= Total score/The number surfaces examine. The minimum score of TMQHPI is 0. The maximum score of TMQHPI is 5.
Saliva sIgA | 0, 4, 5, 9 weeks
  The saliva sIgA level will be evaluated at baseline and different timepoint post-intervention by ELISA.
Halitosis | 0, 4, 5, 9 weeks
  The halitosis will be evaluated at baseline and different timepoint post-intervention by halitosis meter.
Questionnaire assessment | 0, 4, 5, 9 weeks
  The oral health will be evaluated by Oral Health Impact Profile (OHIP) questionnaire. The oral health will be evaluated by Gut Health Assessment questionnaire.The questionnaire is comprised of 26 items.The questionnaire will be evaluated at baseline and different timepoint post-intervention.
Analysis of oral microbiota | 0, 4, 5, 9 weeks
  The change in composition of oral microbiota will be evaluated at baseline and different timepoint post-intervention using real time PCR.

CONTACTS AND LOCATIONS:
Overall Officials: Ju-Hua Wu, PhD, Principal Investigator — Kaohsiung Medical University Chung-Ho Memorial Hospital
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Derived] Lee MK, Chen IH, Hsu IL, Tsai WH, Lee TY, Jhong JH, Liu BC, Huang TY, Lin FK, Chang WW, Wu JH. The impact of Lacticaseibacillus paracasei GMNL-143 toothpaste on gingivitis and oral microbiota in adults: a randomized, double-blind, crossover, placebo-controlled trial. BMC Oral Health. 2024 Apr 20;24(1):477. doi: 10.1186/s12903-024-04251-4. PMID 38643116